CLINICAL TRIAL: NCT05284331
Title: Outcome of Old Patient With Articular With Articular Implant Infection
Acronym: OPWAI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHMS20001
Record Dates: First submitted 2021-09-24; First posted 2022-03-17 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Complications; Implant, Orthopedic, Infection or Inflammation
Keywords: Articular Implant Infection
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- follow-up visit at 6 months and 1 year after inclusion. (Other): addition of a follow-up visit at 6 months and 1 year after inclusion. No treatment will be given specifically for this study. Other visits are part of the normal and usual rhythm of follow-up and evaluation of treatment in these patients
  Interventions: Other: addition of two follow-up visits post infection

INTERVENTIONS:
Other: addition of two follow-up visits post infection — Addition of an additional follow-up visit 6 months post infection and one follow-up visit 1 year post infection.
  No treatment will be given specifically for this study. The change in medical management will only be modified by the addition of these 2 consultations at 6 months and 1 year post infection

SUMMARY:
Articular Implant Infection (AII) is itself a complicated diagnosis and a challenging condition to treat. In elderly patients, the application of existing recommendations is impeded by multiple frailties For a better knowledge of the long-term consequences of AII in elderly patient, the investigators conduct a prospective, multicentric study, whitch aim this is to better evaluate the burden of AII on elderly patients, in terms of quality of life. Secondly, the investigators would like to identify the factors that influence the prognosis, in order to guide further prospective research.

DETAILED DESCRIPTION:
Articular Implant Infection (AII) is itself a complicated diagnosis (diagnosis confirmation, pathogen identification, with appropriate samples) and a challenging condition to treat (long antibiotic exposure, repeated surgery, complex implant change). This condition requires a good cooperation between surgeon and infectious disease specialist, with a comprehension of each one's constraint. In elderly patients, the application of existing recommendations is impeded by multiple frailties (malnutrition, loss of autonomy, polypathology) which make each decision crucial. Indeed, from the choice of surgery to antibiotics management, all medical decision can induce more adverse events than in younger patients. For a better knowledge of the long-term consequences of AII in elderly patient, the investigators conduct a prospective, multicentric study, based on the evaluation of the EQ-5D-5L score during one year after AAI diagnosis in patients older than 75. The investigators evaluate this score and compare different groups of patients, according to age, nutrition status, Charlson comorbidity index, hospital stay length, and loss of autonomy, among others. The aim of this study is to better evaluate the burden of AII on elderly patients, in terms of quality of life. Secondly, the investigators would like to identify the factors that influence the prognosis, in order to guide further prospective research.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized in infectious diseases, surgery, post-emergency unit, or geriatrics,
* diagnosed with a hip or knee prosthesis infection in the previous month according to the SPILF criteria (2009)(1).

Exclusion Criteria:

* Above criteria not met,
* Patient refusal,
* Mild cognitive impairment or more significant.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Changes in the EQ-5D-5L quality of life score | 1 year
  the EQ-5D-5L questionnaire is a European quality of life scale: a first part with questions called "EQ-5D descriptive system" comprising 5 items: mobility, self-care, usual activities, pain and discomfort, anxiety and depression; each item is rated from 1 to 5; 1 corresponding to "no problem", "5" representing "extreme problems or total disability Changes in the EQ-5D-5L quality of life score, 1 year after the onset of symptoms will be evaluated
Changes in the EQ-5D-VAS assessing the patient's general condition, completed by the patient | 1 year
  the EQ-5D-5L questionnaire is completed by a visual analogue scale, called "EQ-5D VAS"; it consists of a 20 cm line, graduated from 0 to 100, where the patient has to indicate how he/she evaluates his/her current state of health, 0 being the worst possible state and 100 the best; Changes in the "EQ-5D VAS" wil be evaluated 1 year after the onset of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: PEJU Martin, Physician, Principal Investigator — Centre Hospitalier Metropole Savoie
Locations (1):
- Centre Hospitalier Métropole Savoie, Chambéry, France